CLINICAL TRIAL: NCT05841693
Title: Quality of Recovery in Parturients Consumed Preoperative Carbohydrate Fluid for Elective Cesarean Delivery- An Obsevational Study
Brief Title: Quality of Recovery in Parturients Consumed Preoperative Carbohydrate Fluid for Elective Cesarean Delivery
Acronym: QoR-10
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Karamanoğlu Mehmetbey University (Other)
Responsible Party: Principal Investigator, Ozlem Dulger, Assist Prof, Karamanoğlu Mehmetbey University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1111
Record Dates: First submitted 2023-04-11; First posted 2023-05-03 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Quality of Life; Breastfeeding; Postoperative Pain; Postoperative Nausea
Keywords: Cesarean Delivery; Quality of Recovery; Preoperative Carbonhyrate Fluid
MeSH Terms: conditions — Breast Feeding; Pain, Postoperative; Postoperative Nausea and Vomiting | interventions — Carbohydrates

STUDY DESIGN:
Intervention Model Description: Randomized, double blinded
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The patients in CHO group will be offered carbohyrate rich preoperative fluid on the other hand the patients in Control Group will be offered placebo fluids resemble to carbohydrate rich preoperative drink. The investigators, care provider and outcome accessors also will be blinded to the group assignment of the patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental ( Carb Group) (Active Comparator): Preoperative education will be provided by researchers to the patients on the ward before fluid intake.Solid food and drinking will be forbidden after 24:00 p.m the day before surgery. The Carb group will consume carbonhydrate fluid two hours before the surgery.
  Interventions: Drug: Carbohydrate
- Standard Care (Non-carb Group) (Placebo Comparator): Preoperative education will be provided by researchers to the patients on the ward before fluid intake. Solid food and drinking will be forbidden after 24:00 p.m the day before surgery.The Non-carb Group will consume same amount of placebo fluid as Carb Group two hours before the surgery
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Carbohydrate — The experimental group of patients will consume the carbohydrate rich fluid 2 hours before the elective CD.
  Other Names: Preoperative carbohydrate rich feeding solution
  Arms: Experimental ( Carb Group)
Drug: Placebo — The control group will be offered same amount of placebo fluid.
  Other Names: Preoperative placebo fluid
  Arms: Standard Care (Non-carb Group)

SUMMARY:
The establishment of the Enhanced Recovery After Cesarean protocols resulted in to the production of specific care pathways with the aim of optimizing recovery after cesarean delivery (CD) and to reduce the costs to the health care system. Carbohydrate rich fluids are offered in this aspect to enhance postoperative quality of recovery. The primary aim of this randomised control trial is to assess the impact of pre-operative carbohydrate loading on obstetric quality of recovery after elective cesarean section.

DETAILED DESCRIPTION:
The 10-item Obstetric Quality-of-Recovery scale is a validated patient-reported outcome questionnaire that evaluates recovery quality after delivery. Carbohydrate loading before the surgery in obstetric patients reduce the incidence of nausea and vomiting and reduce insulin resistance. The shortened pre-operative fasting period, in addition to the positive metabolic effects, enhance the post-operative recovery and shorten the hospital stay. Postoperatively, it is also crucial for the mother to heal rapidly and be able to care for her child on her own. Although a lot of effects of the preoperative carbohydrate loading has been studied yet, the OQR-10 scale and after carbohydrate loading has not been investigated yet.

All mothers undergoing a planned CD in the Karaman Training and Research Hospital will be invited to participate. Mothers will be divided into two groups. One group will receive carbohydrate solution ( Carb Group) and the other will consume same amount of placebo fluid (Noncarb Group).

The aim of this study is to determine the effect of carbonhydrate rich solutions on quality of recovery of parturients undergoing elective CD with Obstetric Quality of Recovery-10 (ObsQoR-10) Scoring Tool.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 years old and over
* Term singleton pregnancy
* Undergoing planned caesarean delivery at Karaman Training and Research Hospital
* Patients who have given informed written consent

Exclusion Criteria:

* Patients who have refused, are unable to give or have withdrawn consent
* Patients with American Society of Anesthesiologists (ASA) classification of 4 or greater
* Patients with history of chronic pain, chronic use of analgesic drugs, or history of opioid or intravenous drug abuse
* Patients who have refused spinal anesthesia, or those in whom it is contraindicated.
* Pregnancy with preeclampsia or eclampsia
* Pregnancy with gestational diabetes mellitus or diabetes mellitus

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female patients undergoing electve cesarean delivery
Enrollment: 100 (Actual)
Dates: Start 2023-05-12 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-03-10 (Actual)

PRIMARY OUTCOMES:
Obstetric Quality of Recovery-10 (ObsQoR-10) score 24 hours | 24 hours
  ObsQoR-10 score at 24 hours after surgery for both parturients consumed carbohydrate rich solution or placebo fluid. There are 10 questions, and the results are tabulated out of 100. The higher the overall score out of 100, the better quality of recovery a patient is experiencing.

SECONDARY OUTCOMES:
Obstetric Quality of Recovery-10 (ObsQoR-10) score 72 hours | 72 hours
  ObsQoR-10 score at 72 hours after surgery for both parturients consumed carbohydrate rich solution or placebo fluid. There are 10 questions, and the results are tabulated out of 100. The higher the overall score out of 100, the better quality of recovery a patient is experiencing.
Obstetric Quality of Recovery-10 (ObsQoR-10) score 7 days | 7 days
  ObsQoR-10 score at 7 days after surgery for both parturients consumed carbohydrate rich solution or placebo fluid. There are 10 questions, and the results are tabulated out of 100. The higher the overall score out of 100, the better quality of recovery a patient is experiencing.
Hospital discharge | 7 days
  The parturients will be discharged from the hospital after they met the discharge criteria. This parameter reported as number of days after the operation to the day in which the patient met discharge criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Ozlem Dulger, Assist Prof, Principal Investigator — Karaman Training and Research Hospital
Locations (1):
- Karaman Training and Research Hospital, Karaman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data of the study will be shared on demand.